CLINICAL TRIAL: NCT04440852
Title: Effect of TEACCH Program on the Rehabilitation Training for Preschool Children With Autistic Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Randomized, Controlled Trial of an Intervention for Preschool Children With Autism: TEACCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Mental Health Centre (Other)
Collaborators: Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2016(53)
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Autism Spectrum Disorder
Keywords: TEACCH
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEACCH intervention (Experimental): TEACCH intervention for ASD
  Interventions: Behavioral: TEACCH
- conventional rehabilitation group (No Intervention): Other conventional interventions

INTERVENTIONS:
Behavioral: TEACCH — The Treatment and Education of Autistic and Communication Handicapped Children
  Arms: TEACCH intervention

SUMMARY:
This study is design to evaluate the efficacy of the Treatment and Education of Autistic and Communication Handicapped Children (TEACCH) on the rehabilitation for preschool children with autism spectrum disorders (ASD) in China.A case-randomized controlled study was conducted.Sixty children diagnosed with ASD between 36 and 90 months of age were randomly assigned to the a TEACCH intervention group or a control group.The control group was subjected to regular rehabilitation training, the TEACCH group carried out TEACCH training besides regular rehabilitation training for 6 months. Chinese Version of Psycho-educational Profile-3rd edition (CPEP-3) was used to evaluate the effectiveness of TEACCH rehabilitation training.

DETAILED DESCRIPTION:
Statistical analysis plan:The results were analyze using descriptive, t-test and ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by two children's psychiatrists above the level of the attending physician, in accordance with the diagnostic criteria of DSM-V (Diagnostic and Statistical Manual of Mental Disorder, fifth revised) children's autism spectrum disorder issued by the United States in 2013. Diagnostic screening scales include Autism Behavior Checklist (ABC), Childhood Autism Rating Scale (CARS), and Modified Checklist for Autism in Toddlers (M-CHAT) (for under 4 years old), Social Communication Questionnaire (SCQ) (for over 4 years old), all children' scores above the scale suggest ASD performance;
* able to cooperate with clinical evaluation and related examinations, and the guardian signs the informed consent to agree to participate in the study.

Exclusion Criteria:

* combined with other mental illnesses such as ADHD, with major physical and nervous system diseases;
* serious self-harm.

Ages: 36 Months to 90 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Chinese Version of Psycho-educational Profile-3rd edition (CPEP-3) | pretest
  a validated assessment tool that comprehensively measures the development of Chinese children with ASD
Chinese Version of Psycho-educational Profile-3rd edition (CPEP-3) | posttest: 6 months to pretest
  a validated assessment tool that comprehensively measures the development of Chinese children with ASD
Chinese Version of Psycho-educational Profile-3rd edition (CPEP-3) | 6 months follow-up : 1 year to pretest
  a validated assessment tool that comprehensively measures the development of Chinese children with ASD

CONTACTS AND LOCATIONS:
Overall Officials: Hongling Zeng, Master, Study Director — Wuhan Mental Health Centre
Locations (1):
- Wuhan Mental Health Centre, Wuhan, Hubei, China